CLINICAL TRIAL: NCT07248761
Title: Efficacy of Early Administration of Hydrocortisone in Shock in Preterm Neonates of Less Than 1,500 g
Brief Title: Early Hydrocortisone Versus Regular Treatment in Shock in Extremely Preterm Neonates - an Open Randomized Controlled Trial
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2024-3606-155
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-06

CONDITIONS: Shock; Preterm Birth Complication; Preterm Intraventricular Hemorrhage; Asphyxia Perinatal; Distress Respiratory Syndrome; Hyperglycaemia (Non Diabetic); Neonatal Sepsis, Early-Onset; Neonatal Sepsis, Late-Onset; NEC - Necrotizing Enterocolitis; Patent Ductus Arteriosus in Preterm Infants; Intestinal Perforation
Keywords: Preterm neonates; Shock; Treatment; Hydrocortisone; Early
MeSH Terms: conditions — Shock; Pulmonary Atelectasis; Hyperglycemia; Neonatal Sepsis; Enterocolitis, Necrotizing; Intestinal Perforation

STUDY DESIGN:
Intervention Model Description: The regular group will receive the treatment for shock according to their attending neonatologist. The experimental group will receive the same treatment plus Hydrocortisone parallel to the first vasoactive drug.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm neonates in shock who receive regular treatment. (Active Comparator): The treatment this group receives is determined by the attending neonatologist. It may o may not include Hydrocortisone at some point of the evolution of the disease.
  Interventions: Other: Vasoactive drug therapies
- Preterm neonates in shock who receive regular treatment plus Hydrocortisone from the beginning. (Experimental): This group receives the treatment that the attending neonatologist determines plus Hydrocortisone since the initiation of vasoactive drugs.
  Interventions: Drug: Intravascular Hydrocortisone (stress dosage): 1 mg/k/dose each 8 hours for 5 days

INTERVENTIONS:
Drug: Intravascular Hydrocortisone (stress dosage): 1 mg/k/dose each 8 hours for 5 days — The "Early Hydrocortisone Group" will be receiving Hydrocortisone since the diagnosis of shock and the vasoactive drugs are initiated.
  Arms: Preterm neonates in shock who receive regular treatment plus Hydrocortisone from the beginning.
Other: Vasoactive drug therapies — This group will receive the treatment that the attending physician will decide. It may include any kind of vasoactive drug and, at some point, Hydrocortisone if the attending considers the patient is going through a "Vasoactive resistant shock".
  Arms: Preterm neonates in shock who receive regular treatment.

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of early use of hydrocortisone (since the diagnosis of shock) for its resolution within the first 72 hours in premature infants under 1,500 g. The main questions it aims to answer are:

* Does the early use of hydrocortisone help solve shock in preterm infants under 1500 g faster than the standard treatment?
* Does the early use of hydrocortisone help prevent death within the first seven days of presentation of shock in comparison to premature infants who receive regular treatment?

Researchers will compare the early use of hydrocortisone plus the standard treatment to solve shock against just standard treatment.

Participants will:

* Be randomized to receive standard treatment for shock according to their neonatologist or this standard treatment plus hydrocortisone as soon as the diagnosis is done and treatment is started.
* Be followed either until shock is solved or if they present death due to this event of shock.

DETAILED DESCRIPTION:
WORK STRATEGY:

PHASE I:

1. Initially, the main investigators carried out an information campaign aimed at neonatologists in the Neonatal Intensive Care Unit to unify criteria on the diagnosis of shock, provide information on current developments in treatment of premature newborns, and publicize the characteristics of the research project.

   1. A shock algorithm was developed according to the most recent evidence-based recommendations to unify criteria for the diagnosis of shock in premature infants and its treatment according to the pathophysiology.
   2. The algorithm is available on the computers of each of the physicians in the NICU.
   3. The algorithm has been disseminated to all physicians through several talks during their shift.
   4. This algorithm was also printed on 1.5 x 2 meter posters, which were placed in the NICU physicians' offices for quick access.
   5. All physicians have been invited to collaborate on the research project.
2. On the other hand, an information campaign has been carried out aimed at the nursing staff of the NICU with the aim of updating their knowledge on the correct measurement of blood pressure in premature newborns and unifying criteria.

   1. Posters were made with updated information on blood pressure measurement.
   2. These posters were printed on 1.2 x 70 cm sheets. The posters were placed in strategic locations in the NICU so that the information was readily available to staff.
   3. An informative talk was given to the nursing staff of both services and all three shifts about the research project and the importance of their participation in the early detection of shock symptoms.

PHASE II:

1. The investigators identify very low birth weight subjects (<1,500 g) who enter the NICU.
2. After the subjects are admitted, the investigators explain to their parents that they may participate in this clinical trial if their children present clinical deterioration during the first 14 days of hospitalization. They are given a detailed explanation of shock, standard treatment, the use of hydrocortisone, its benefits, and potential risks. If the parents agree to their children participating in the trial, the attending physician has them read and sign the informed consent form.
3. Subjects with informed parental consent are followed up during the first 14 days of extrauterine life to include in the study those diagnosed with shock:

   1. The diagnosis of shock is made by the attending physician, confirming the clinical data with the nursing staff.
   2. Both the doctor and the nursing staff record the clinical data found in their respective notes.
4. When the attending physician decides to initiate aminergic support, he or she should take a randomization form, which is located in a box within reach of the physician's office:

   1. Block randomization is performed by a research associate blinded to the identity of the subjects in blocks of 5 using a random number generator table based on Stata 13. The objective of this randomized sampling is to estimate the effects of the treatments and the blocks and to test the hypothesis that all levels of the main factor produce the same effect, versus the alternative that at least two differ significantly. These randomized blocks are placed in a box with the corresponding treatment so that the attending physicians can take a paper with the corresponding assignment.
   2. All neonatologists have been informed about the ongoing study and the presence of a "randomization" box with papers inside. Two types of papers have been placed in the box, depending on the corresponding randomization. The papers may have two legends: one consisting of "Standardized treatment (standard treatment according to the criteria of the attending physician)" and the other "Standardized treatment plus hydrocortisone (1 mg/kg/day every 8 hours)."
   3. The attending physician will establish in the medical note and inform the nursing staff the type of treatment the subject will receive, whether the usual treatment or the usual treatment plus early hydrocortisone. The nursing staff has been instructed that if the subject is randomized to the second group, they should begin administering and preparing both the vasoactive amines and hydrocortisone as soon as possible.
5. At the start of treatment in both groups, the cardiologist will perform an initial echocardiographic evaluation using the Vivid 4 device with a 6 MHz sector transducer. The evaluation is a protocol used to exclude congenital cardiac malformations and assess both cardiac function and hemodynamic characteristics. The evaluation includes the following:

   1. Windows: Sites where the transducer is placed to obtain specific measurements. These include the subcostal short and long axis, the parasternal short and long axis, the apical window, and the suprasternal window.
   2. Measurements: All valves, pulmonary branches, aortic arch, and all four chambers.
   3. Pulmonary and systemic venous return should be defined, as well as the shunts present and ventricular function (systolic and diastolic).
   4. If a patent ductus arteriosus is found, the following will be evaluated:

   i. Duct characteristics: duct diameter, short circuit and flow through the duct.

   ii. Diastolic flow of the Middle Cerebral Artery (MCA): the transducer is placed in a plane transverse to the coronal suture, the MCA is identified using color Doppler and the systolic and diastolic flow pattern is observed in M mode to determine if there is diastolic steal, that is, if there is absent or reverse diastolic flow (see Figure 3.).

   iii. Diastolic flow in the celiac trunk and superior mesenteric artery: by placing the probe in the subcostal window, color Doppler is used to locate the arteries and then M-mode flow is obtained to assess flow during systole and diastole. This identifies any flow disturbances during diastole (see Figure 4).
6. After starting vasoactive agents, close monitoring of vital signs and clinical progress of each patient will be carried out using nursing sheets and medical notes (electronic and physical records):

   A) The vital signs recorded by the nurse will be those taken from the electronic monitor. Specifically, blood pressure will be measured noninvasively, using the Mindray-Bene View T5 system, as well as width-appropriate cuffs.

   B) Aminergic support used, time of use and dose. C) Associated comorbidities that are diagnosed. D) Type of supplemental oxygen support (assisted mechanical ventilation, CPAP, or free-flow oxygen) and its duration.
7. Subjects will be followed up for seven days after the start of treatment.
8. The variables of interest will be collected on the collection sheet.
9. A database will be generated with the collected information, which will be analyzed using Stata version 13.

BIOSECURITY MEASURES:

Patient safety is a priority for health systems worldwide. Through the Global Partnership for Patient Safety, the World Health Organization (WHO) established the goal of preventing adverse events during care in health institutions, thus ensuring risk-free care.

Individuals in the neonatal stage of development are more vulnerable to injury during their hospital stay, so specific safety measures are needed to prevent risks during their care. Accordingly, guidelines have been proposed for this age group, based on the six International Patient Safety Goals established by the World Health Organization (WHO). To minimize the possibility of adverse events occurring during the care of study subjects, researchers and collaborators ensure the following:

1. Correctly identify subjects before randomization and throughout the trial by providing full name, social security number, date of birth, and study participant folio number.
2. Improved effective communication through verification of the indication of the group to which it belongs (control vs. intervention) by two people verbally and in writing, that is, by the researcher in charge and the assigned physician.
3. Improving the safety of high-risk medications: Although hydrocortisone is not considered a high-risk medication as such, it must be administered correctly, ensuring that the prescription is 1 milligram per kilogram of the subject's weight every 8 hours, as directed by the nursing staff. Both the principal investigator and the attending physician must verify that the prescription is correctly written and understandable to the nursing staff.
4. Ensuring surgeries are performed in the right location, with the right procedure and with the right patient: routine NICU activities.
5. Reduction of healthcare-acquired infections: Continuous monitoring for the presence of opportunistic sepsis, especially Candida sp., should be carried out. If it is present in more than 20%, the trial should be stopped.
6. Reducing the risk of patient injuries from falls: Routine NICU activities.

In addition, the following points will be considered to ensure the safety of newborns in this clinical trial:

* First of all, the patient must meet a series of conditions, the so-called inclusion criteria and exclusion criteria.
* Informed consent: Parents must give their permission for the subject to participate in the study after receiving an explanation about the study and reading the informed consent form, speaking with their treating physician and the principal investigator, and asking questions. Once the subject has been selected, parents or guardians must be aware of and informed about the characteristics of the study. The information is provided in writing and is written in clear and understandable terms. Furthermore, the family has the opportunity to receive oral information about any information they do not understand or require clarification. After receiving the information, they are offered a reflection period by those responsible for the study to decide whether to participate and give their free, voluntary, and informed consent by signing the corresponding document. In any case, the researcher accepts the explicit wish of the parents or guardians to refuse to participate in the trial or to withdraw at any time.
* The legal framework establishes the legal procedures and control systems from the start to the end of the clinical trial. Of particular note is NOM-012-SSA3-2012, which establishes the criteria for the execution of health research projects in human subjects. It incorporates, as key safeguards, the protection of minors' rights and the need for experts with training or experience in dealing with minors to participate in the evaluation of clinical trials.
* The clinical trial was initiated until a favorable opinion was obtained from the HGO 4 Research Ethics Committee.
* Data and Safety Monitoring Committee (Interim Analysis): This committee is co-composed of two expert research associates located outside the unit and who receive information from the study subjects to perform a preliminary statistical analysis. These research associates are blinded to patient randomization. They review the study results and may stop the trial if the experimental treatment is causing harm to participants, i.e., if patients in the intervention group have a higher incidence of intestinal perforation than described in the literature (>1.1% in newborns weighing more than 1,000 g up to 1,500 g and >7.4% in newborns weighing less than 1,000 g) or a higher incidence of Candida sp infection (>20%). If a higher incidence of these serious adverse events is observed in the intervention group compared to the control group (statistically and clinically significant), the study will be stopped.
* Upon completion of the study, the researchers agree to publish the results obtained in scientific journals, whether favorable or unfavorable to the working hypothesis. The anonymity of the participating patients will always be maintained.
* The clinical trial was designed to minimize risk to participants, based on an extensive and exhaustive review of the literature on the subject. It is believed that the study subjects do not run any additional risk by participating in the trial; on the contrary, they are more likely to improve their survival and reduce the risk of developing comorbidities associated with shock.
* In this study, it was decided not to use a placebo so that subjects would not be deprived of a treatment necessary for their health. Furthermore, the treating physician will have the option of stopping the administration of hydrocortisone if he or she deems it unsafe for their patient.
* Hydrocortisone dose: The dose of hydrocortisone used is equivalent to the cortisol produced by humans during periods of stress, and the dose with which a lower incidence of side effects has been observed in other clinical trials. The duration of use depends on the subject's clinical course; that is, if the subject's shock resolves within 72 hours and no longer requires aminergic support, hydrocortisone use can be discontinued, allowing subjects to receive this treatment for three to five days. This treatment should not be used for more than five days, as described in the literature.

DATA ANALYSIS:

All randomized subjects will be included in an intention-to-treat analysis. The following data analysis will be performed:

Descriptive statistics: Qualitative variables will be expressed as frequencies and percentages; for quantitative variables, a test will be performed to determine the parametric distribution of the data. Based on the distribution type, these variables will be expressed in measures of central tendency (mean, median) and dispersion (standard deviation, minimum-maximum interval, or interquartile ranges).

If differences are found between treatment groups, an unadjusted analysis and another adjusted for the variable that unbalanced the groups will be performed.

Inferential statistics: By creating comparison groups between subjects with and without early administration of Hydrocortisone, the following analysis will be performed:

1. Bivariate: For qualitative variables, the chi-square or Fisher exact test will be used; for quantitative variables, the Mann-Whitney T or U test will be used. A p-value <0.5 will be considered statistically significant.
2. Outcomes or adverse events will be analyzed using analysis of variance or covariance for continuous outcomes and logistic regression analysis or Fisher's exact test for binary outcomes.
3. The risk difference (RRR) between the two groups with respect to the control and the absolute risk reduction (RAR) will be calculated.
4. Kaplan-Meier curves will be performed to analyze the occurrence of events and the effect of interventions on these events will be evaluated using the Cox proportional hazard model (post-hoc analysis).

ETHICAL ASPECTS:

1. The researcher guarantees that this study complies with the legislation and regulations of Mexico´s General Health Law on Health Research , which provides greater protection to the subjects of the study.
2. In accordance with Article 17 of the Regulations of the General Health Law on Health Research, this project is considered "research with greater than minimum risk," since a clinical intervention is carried out in which Hydrocortisone is administered at physiological doses together with vasoactive amines to very low birth weight newborns diagnosed with Shock.
3. The procedures of this study adhere to the ethical standards, the Regulations of the General Health Law on Research and will be carried out in full compliance with the following principles of the "Declaration of Helsinki" (and its amendments in Tokyo, Venice, Hong Kong and South Africa) where the researcher guarantees that:

   1. A thorough search of the scientific literature on the topic to be addressed was conducted, and the search for new information continues throughout the course of the study.
   2. All study subjects receive standard treatment for septic shock as stipulated in internationally endorsed clinical practice guidelines.
   3. This protocol was reviewed and approved by the Research Ethics Committee and the Local Health Research Committee of the UMAE HGO 4 "Luis Castelazo Ayala" of the Mexican Social Security Institute. The protocol has the following registration number: R-2024-3606-155.
   4. This protocol is carried out by scientifically qualified individuals under the supervision of a team of clinically competent physicians certified in their specialty.
   5. This protocol will maintain the confidentiality of individuals.
   6. This study requires a written informed consent letter. Informed consent is obtained by the subject's attending physician, who is not part of the research associates and who takes special care to ensure that legal guardians are not pressured into participating in the study. Should parents have further questions and require further explanation of the procedures, risks, and benefits, further explanation will be provided by the researcher or a research associate.
4. The principles contained in the Nuremberg Code and the Belmont Report are fully respected.
5. The procedure for inviting participants and obtaining informed consent is as follows: once the birth of a premature infant weighing <1,500 g is registered, the legal guardian(s) will be informed about the possibility of presenting signs of shock and requiring management with amines. They are invited to participate in the research project where they are randomized to receive standard treatment or standard treatment plus early hydrocortisone at physiological doses for three to five days.
6. The procedure for ensuring the confidentiality of personal data and information obtained is as follows: each newborn is assigned a folio consisting of the first letter of the maternal surname and a consecutive number, while the newborn's name and affiliation will remain in custody and password-protected on the computer equipment of the researcher in charge.
7. The guidelines of Good Clinical Practices are followed as a standard for developing this research project. The principal investigator is responsible for monitoring compliance with these guidelines, respect for local laws, and adherence to the protocol. A team has been organized to help meet expectations regarding the number of subjects recruited, the timeframe for recruitment, and the quality of the data generated.
8. Finally, as previously mentioned in the "Biosafety Measures" section, a safety committee has been formed with two associate researchers (blinded to subject randomization) that is conducting an interim analysis to assess whether there is a higher incidence of intestinal perforation or Candida sp. infection than described in the literature in this age group in subjects to whom hydrocortisone is administered early, leading to the discontinuation of this study.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies of 1,500 g or less
* Diagnosis of shock by attending physician during their first 14 days of life

Exclusion Criteria:

* Major physical malformations that compromise life itself.
* Preterm newborns with probable Congenital Adrenal Hyperplasia

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Shock resolution | 72 hours
  The patient is hemodynamically stable and no longer requires vasoactive support.

SECONDARY OUTCOMES:
Mortality. | Seven days.
  The patient does not die secondarily to shock.

CONTACTS AND LOCATIONS:
Overall Officials: ELISA DORANTES ACOSTA, PH D HEALTH SCIENCES, Study Director — Hospital Infantil de Mexico Federico Gomez; EDITH VALDEZ MARTINEZ, PH D MEDICAL ETHICS, Study Director — Unidad de Investigación Médica en Epidemiología Clínica, UMAE Hospital de Pediatría, CMN SXXI, IMSS; HORACIO MARQUEZ GONZALEZ, PH D HEALTH SCIENCES, Study Chair — Unidad de investigación, Hospital Infantil de México Federico Gómez / Cardiopatías Congénitas, UMAE Hospital de Cardiología, CMN SXXI, IMSS.; ADRIANA APOLONIO, MARTINEZ, Study Chair — Servicio de Cardiología Pediátrica y Perinatal de la UMAE HGO4, IMSS; MARIA DEL CARMEN JIMENEZ MARTINEZ, PH D IMMUNOLOGY, Study Chair — POSGRADO EN CIENCIAS MÉDICAS DE LA FACULTAD DE MEDICINA DE LA UNAM; FLOR DE MARIA GRANADOS CANSECO, MASTER´S D HEALTH SCIENCES, Principal Investigator — UMAE, HOSPITAL DE GINECO-OBSTETRICIA NO. 4 "LUIS CASTELAZO AYALA", IMSS
Locations (1):
- UMAE Hospital de Gineco Obstetricia No. 4 "Luis Castelazo Ayala", IMSS, Mexico City, ALVARO OBREGON, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared accordingly to the variables taken into account in this study. The epidemiological information and relevant clinical information will be shared but the identification of the individuals will be enclosed for ethical purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Unending.
Access Criteria: Pediatricians, Neonatologists, Cardiologists, Intensive Care Pediatricians Epidemiological variables / Clinical variables / Outcomes All statistical analyses will be available if asked for by e-mail. Every investigator already included will be able to review requests via electronic mail.

REFERENCES:
- [Background] Patra K, Greene MM, Silvestri JM. Neurodevelopmental impact of hydrocortisone exposure in extremely low birth weight infants: outcomes at 1 and 2 years. J Perinatol. 2015 Jan;35(1):77-81. doi: 10.1038/jp.2014.133. Epub 2014 Jul 31. PMID 25078865
- [Background] Rademaker KJ, Uiterwaal CS, Groenendaal F, Venema MM, van Bel F, Beek FJ, van Haastert IC, Grobbee DE, de Vries LS. Neonatal hydrocortisone treatment: neurodevelopmental outcome and MRI at school age in preterm-born children. J Pediatr. 2007 Apr;150(4):351-7. doi: 10.1016/j.jpeds.2006.10.051. PMID 17382109
- [Background] Baud O, Maury L, Lebail F, Ramful D, El Moussawi F, Nicaise C, Zupan-Simunek V, Coursol A, Beuchee A, Bolot P, Andrini P, Mohamed D, Alberti C; PREMILOC trial study group. Effect of early low-dose hydrocortisone on survival without bronchopulmonary dysplasia in extremely preterm infants (PREMILOC): a double-blind, placebo-controlled, multicentre, randomised trial. Lancet. 2016 Apr 30;387(10030):1827-36. doi: 10.1016/S0140-6736(16)00202-6. Epub 2016 Feb 23. PMID 26916176
- [Background] Ramaswamy VV, Kumar G, Pullattayil S AK, Aradhya AS, Suryawanshi P, Sahni M, Khurana S, Saini SS, K R, Dhir SK, Chawla D, Kumar P, More K. Timing of hydrocortisone therapy in neonates with shock: a systematic review, meta-analysis, and clinical practice guideline. Front Pediatr. 2025 Mar 12;13:1491976. doi: 10.3389/fped.2025.1491976. eCollection 2025. PMID 40144277
- [Background] Kumbhat N, Noori S. Corticosteroids for Neonatal Hypotension. Clin Perinatol. 2020 Sep;47(3):549-562. doi: 10.1016/j.clp.2020.05.015. Epub 2020 May 22. PMID 32713450
- [Background] Agakidou E, Chatziioannidis I, Kontou A, Stathopoulou T, Chotas W, Sarafidis K. An Update on Pharmacologic Management of Neonatal Hypotension: When, Why, and Which Medication. Children (Basel). 2024 Apr 19;11(4):490. doi: 10.3390/children11040490. PMID 38671707
- [Background] Dudeja S, Saini SS, Sundaram V, Dutta S, Sachdeva N, Kumar P. Early hydrocortisone verses placebo in neonatal shock- a double blind Randomized controlled trial. J Perinatol. 2025 Mar;45(3):342-349. doi: 10.1038/s41372-025-02222-3. Epub 2025 Feb 13. PMID 39948354
- [Background] Watterberg KL, Shaffer ML, Mishefske MJ, Leach CL, Mammel MC, Couser RJ, Abbasi S, Cole CH, Aucott SW, Thilo EH, Rozycki HJ, Lacy CB. Growth and neurodevelopmental outcomes after early low-dose hydrocortisone treatment in extremely low birth weight infants. Pediatrics. 2007 Jul;120(1):40-8. doi: 10.1542/peds.2006-3158. PMID 17606560
- [Background] Watterberg KL. Hydrocortisone Dosing for Hypotension in Newborn Infants: Less Is More. J Pediatr. 2016 Jul;174:23-26.e1. doi: 10.1016/j.jpeds.2016.04.005. Epub 2016 May 4. No abstract available. PMID 27156187
- [Background] Ng PC, Lee CH, Bnur FL, Chan IH, Lee AW, Wong E, Chan HB, Lam CW, Lee BS, Fok TF. A double-blind, randomized, controlled study of a "stress dose" of hydrocortisone for rescue treatment of refractory hypotension in preterm infants. Pediatrics. 2006 Feb;117(2):367-75. doi: 10.1542/peds.2005-0869. PMID 16452355
- [Background] Altit G, Vigny-Pau M, Barrington K, Dorval VG, Lapointe A. Corticosteroid Therapy in Neonatal Septic Shock-Do We Prevent Death? Am J Perinatol. 2018 Jan;35(2):146-151. doi: 10.1055/s-0037-1606188. Epub 2017 Aug 24. PMID 28838003
- [Background] Higgins S, Friedlich P, Seri I. Hydrocortisone for hypotension and vasopressor dependence in preterm neonates: a meta-analysis. J Perinatol. 2010 Jun;30(6):373-8. doi: 10.1038/jp.2009.126. Epub 2009 Aug 20. PMID 19693023
- [Background] Subhedar NV, Duffy K, Ibrahim H. Corticosteroids for treating hypotension in preterm infants. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD003662. doi: 10.1002/14651858.CD003662.pub3. PMID 17253493
- [Background] Noori S, Friedlich P, Wong P, Ebrahimi M, Siassi B, Seri I. Hemodynamic changes after low-dosage hydrocortisone administration in vasopressor-treated preterm and term neonates. Pediatrics. 2006 Oct;118(4):1456-66. doi: 10.1542/peds.2006-0661. PMID 17015536
- [Background] Ng PC, Lam CW, Fok TF, Lee CH, Ma KC, Chan IH, Wong E. Refractory hypotension in preterm infants with adrenocortical insufficiency. Arch Dis Child Fetal Neonatal Ed. 2001 Mar;84(2):F122-4. doi: 10.1136/fn.84.2.f122. PMID 11207229
- [Background] Efird MM, Heerens AT, Gordon PV, Bose CL, Young DA. A randomized-controlled trial of prophylactic hydrocortisone supplementation for the prevention of hypotension in extremely low birth weight infants. J Perinatol. 2005 Feb;25(2):119-24. doi: 10.1038/sj.jp.7211193. PMID 15329742
- [Background] Salas G, Travaglianti M, Leone A, Couceiro C, Rodriguez S, Farina D. [Hydrocortisone for the treatment of refractory hypotension: a randomized controlled trial]. An Pediatr (Barc). 2014 Jun;80(6):387-93. doi: 10.1016/j.anpedi.2013.08.004. Epub 2013 Oct 16. Spanish. PMID 24139558
- [Background] Morabito LA, Corica D, Pepe G, Li Pomi A, Aversa T, Wasniewska MG. Critical illness-related corticosteroid insufficiency (CIRCI) in paediatric patients: a diagnostic and therapeutic challenge. Ital J Pediatr. 2024 Mar 11;50(1):46. doi: 10.1186/s13052-024-01616-x. PMID 38462639
- [Background] Rulli I, Carcione AM, D'Amico F, Quartarone G, Chimenz R, Gitto E. Corticosteroids in Pediatric Septic Shock: A Narrative Review. J Pers Med. 2024 Dec 17;14(12):1155. doi: 10.3390/jpm14121155. PMID 39728068
- [Background] Schlapbach LJ, Watson RS, Sorce LR, Argent AC, Menon K, Hall MW, Akech S, Albers DJ, Alpern ER, Balamuth F, Bembea M, Biban P, Carrol ED, Chiotos K, Chisti MJ, DeWitt PE, Evans I, Flauzino de Oliveira C, Horvat CM, Inwald D, Ishimine P, Jaramillo-Bustamante JC, Levin M, Lodha R, Martin B, Nadel S, Nakagawa S, Peters MJ, Randolph AG, Ranjit S, Rebull MN, Russell S, Scott HF, de Souza DC, Tissieres P, Weiss SL, Wiens MO, Wynn JL, Kissoon N, Zimmerman JJ, Sanchez-Pinto LN, Bennett TD; Society of Critical Care Medicine Pediatric Sepsis Definition Task Force. International Consensus Criteria for Pediatric Sepsis and Septic Shock. JAMA. 2024 Feb 27;331(8):665-674. doi: 10.1001/jama.2024.0179. PMID 38245889
- [Background] Schwarz CE, Dempsey EM. Management of Neonatal Hypotension and Shock. Semin Fetal Neonatal Med. 2020 Oct;25(5):101121. doi: 10.1016/j.siny.2020.101121. Epub 2020 May 21. PMID 32473881
- [Background] Ng PC, Lam CW, Lee CH, Ma KC, Fok TF, Chan IH, Wong E. Reference ranges and factors affecting the human corticotropin-releasing hormone test in preterm, very low birth weight infants. J Clin Endocrinol Metab. 2002 Oct;87(10):4621-8. doi: 10.1210/jc.2001-011620. PMID 12364445
- [Background] Ng PC, Lee CH, Lam CW, Ma KC, Fok TF, Chan IH, Wong E. Transient adrenocortical insufficiency of prematurity and systemic hypotension in very low birthweight infants. Arch Dis Child Fetal Neonatal Ed. 2004 Mar;89(2):F119-26. doi: 10.1136/adc.2002.021972. PMID 14977894
- [Background] van de Loo M, van Kaam A, Offringa M, Doyle LW, Cooper C, Onland W. Corticosteroids for the prevention and treatment of bronchopulmonary dysplasia: an overview of systematic reviews. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD013271. doi: 10.1002/14651858.CD013271.pub2. PMID 38597338
- [Background] Baud O, Torchin H, Butin M, Flamant C, Nuytten A. Prophylactic low-dose hydrocortisone in neonates born extremely preterm: current knowledge and future challenges. Pediatr Res. 2025 Jul;98(1):65-71. doi: 10.1038/s41390-024-03756-6. Epub 2024 Nov 26. PMID 39592771
- [Background] Ng PC, Wong SP, Chan IH, Lam HS, Lee CH, Lam CW. A prospective longitudinal study to estimate the "adjusted cortisol percentile" in preterm infants. Pediatr Res. 2011 Jun;69(6):511-6. doi: 10.1203/PDR.0b013e31821764b1. PMID 21364494
- [Background] Baud O, Watterberg KL. Prophylactic postnatal corticosteroids: Early hydrocortisone. Semin Fetal Neonatal Med. 2019 Jun;24(3):202-206. doi: 10.1016/j.siny.2019.04.007. Epub 2019 Apr 20. PMID 31043325
- [Background] Huysman MW, Hokken-Koelega AC, De Ridder MA, Sauer PJ. Adrenal function in sick very preterm infants. Pediatr Res. 2000 Nov;48(5):629-33. doi: 10.1203/00006450-200011000-00013. PMID 11044483
- [Background] Quintos JB, Boney CM. Transient adrenal insufficiency in the premature newborn. Curr Opin Endocrinol Diabetes Obes. 2010 Feb;17(1):8-12. doi: 10.1097/MED.0b013e32833363cc. PMID 19881342
- [Background] Kharrat A, Diambomba Y, Jain A. Corticosteroid use in neonatal hypotension: A survey of Canadian neonatologists. Pediatr Neonatol. 2024 Sep;65(5):451-456. doi: 10.1016/j.pedneo.2023.09.013. Epub 2024 Feb 5. PMID 38388227
- [Background] Ng PC. Adrenocortical insufficiency and refractory hypotension in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2016 Nov;101(6):F571-F576. doi: 10.1136/archdischild-2016-311289. Epub 2016 Sep 6. PMID 27601464
- [Background] Spaggiari V, Passini E, Crestani S, Roversi MF, Bedetti L, Rossi K, Lucaccioni L, Baraldi C, Della Casa Muttini E, Lugli L, Iughetti L, Berardi A. Neonatal septic shock, a focus on first line interventions. Acta Biomed. 2022 Jul 1;93(3):e2022141. doi: 10.23750/abm.v93i3.12577. PMID 35775767
- [Background] Saini SS, Shrivastav AK, Kumar J, Sundaram V, Mukhopadhyay K, Dutta S, Ray P, Kumar P. Predictors of Mortality in Neonatal Shock: A Retrospective Cohort Study. Shock. 2022 Feb 1;57(2):199-204. doi: 10.1097/SHK.0000000000001887. PMID 34798634
- [Background] Seri I, Noori S. Diagnosis and treatment of neonatal hypotension outside the transitional period. Early Hum Dev. 2005 May;81(5):405-11. doi: 10.1016/j.earlhumdev.2005.03.008. PMID 15882935
- [Background] Bhat BV, Plakkal N. Management of Shock in Neonates. Indian J Pediatr. 2015 Oct;82(10):923-9. doi: 10.1007/s12098-015-1758-7. Epub 2015 May 21. PMID 25990594
- [Background] Mullaly R, El-Khuffash AF. Haemodynamic assessment and management of hypotension in the preterm. Arch Dis Child Fetal Neonatal Ed. 2024 Feb 19;109(2):120-127. doi: 10.1136/archdischild-2022-324935. PMID 37173119
- [Background] Cayabyab R, McLean CW, Seri I. Definition of hypotension and assessment of hemodynamics in the preterm neonate. J Perinatol. 2009 May;29 Suppl 2:S58-62. doi: 10.1038/jp.2009.29. PMID 19399011
- [Background] Wu TW, Noori S. Recognition and management of neonatal hemodynamic compromise. Pediatr Neonatol. 2021 Feb;62 Suppl 1:S22-S29. doi: 10.1016/j.pedneo.2020.12.007. Epub 2020 Dec 24. PMID 33485823
- [Background] Johnson PJ. Hydrocortisone for Treatment of Hypotension in the Newborn. Neonatal Netw. 2015;34(1):46-51. doi: 10.1891/0730-0832.34.1.46. PMID 26803045
- [Background] Barrington KJ. Hypotension and shock in the preterm infant. Semin Fetal Neonatal Med. 2008 Feb;13(1):16-23. doi: 10.1016/j.siny.2007.09.002. Epub 2007 Oct 31. PMID 17974512